CLINICAL TRIAL: NCT07085351
Title: Developing EEG Biomarkers for OUD Diagnostic, Prognostic, and Predictive Purposes
Brief Title: EEG Biomarkers for OUD: Diagnostic, Prognostic, and Predictive Applications
Status: Recruiting | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ciro Ramos Estebanez, Principal Investigator, University of Illinois at Chicago
Other Study IDs: STUDY2023-1092; R43DA058979 (NIH)
Record Dates: First submitted 2025-07-08; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Opiod Use Disorder
Keywords: opioid use disorder; EEG
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Opioid Use Disorder: Diagnosed Opioid Use Disorder subjects will perform 2 EEG sessions done at the initial visit and one week later. EEG recordings will be taken to monitor brain activity
- Healthy Control: Age-matched healthy controls. Subjects will perform 2 EEG sessions done at the initial visit and one week later. EEG recordings will be taken to monitor brain activity

SUMMARY:
The US is suffering from a national opioid epidemic characterized by significant costs, overdoses, and deaths. Conventional Opioid Use Disorder (OUD) treatments (i.e., pharmacological and psychosocial interventions) are characterized by limited or diminishing efficacy, ceiling effects, and/or serious side effects. The availability of validated OUD biomarkers would be a key step in the development and approval of better treatments. Ultimately, the scarcity of OUD biomarkers represents a significant unmet need in the fight against opioid addiction as recognized by NIDA and the FDA with their support for development of Medical Device Development Tools (MDDT) and biomarker tests for OUD. Advances in neuroimaging techniques, and in particular recent evidence supports electroencephalography (EEG) as a promising candidate to investigate the correlation between addiction and brain state. To address the clear medical and market need for OUD biomarkers, this is a feasibility study to identify and assess potential EEG biomarkers for OUD diagnoses, disease monitoring, and prediction of OUD treatment response.

DETAILED DESCRIPTION:
We will recruit up to 130 subjects for this study, with the intention of enrolling 50 OUD subjects at various stages of treatment and 20 age-matched non-OUD controls.

Eligible subjects will contact or give verbal permission to be contacted via their referring provider, by a co-investigator to obtain more information about the study. At the first point of contact (usually a phone call), study co- investigator will administer a phone-screening questionnaire. Once the phone screening process is complete, the information gathered by the co-investigator will be taken to the PI of the study for further review to confirm eligibility. Data obtained from screening will be safely stored in the PI's locked office.

Informed consent will be obtained by the study PI and/or a co-investigator (not involved in the patient's care) in person. The test procedures will be described and the testing equipment will be shown to the subject. Study co-investigators will clearly explain all the procedures and risks of the testing outlined in the consent form. The subject will be given the time needed to consider their decision and will be encouraged to ask questions, both during the initial phone interview and throughout the study. The PI or a co-investigator will answer any questions regarding the study at the time consent is given. Once enrolled, the subject may pause or terminate his/her participation at any time during the study.

Procedures Involved* This is an observational study that includes an EEG at rest and also an EEG conducted while the subject is simultaneously completing a computer assessment. The study will have 50 OUD patients and 20 age-matched controls. Subjects will undergo EEG testing in addition to testing done concurrently with computer assessments. An additional visit will be conducted around 1 week after the initial visit. Additionally, subjects will undergo questionnaires/assessments regarding demographics, HPI, craving, mood, impulsivity, and drug use. Urine toxicology and Hair follicle (when available) will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* For OUD Subjects:

  1. Providing informed consent to participate in the study.
  2. 22 to 85 years old.

Having a diagnosis of OUD

• OUD of more than 6 months duration as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM-5) [71] with a positive urine toxicology screen who still feel craving.

4. Lives in immediate area with no plans to relocate.

For age-matched controls:

1. Providing informed consent to participate in the study.
2. 22 to 85 years old.
3. Lives in immediate area with no plans to relocate

Exclusion Criteria:

* For OUD Subjects:

  1. Recently started on antiepileptic drug therapy.
  2. Ingestion of poppy seeds or herbal teas containing Papaveris fructus (may cause a positive opiate test for morphine, codeine [72,73]).
  3. History of neurological disorders involving stroke, brain tumors, or epilepsy as self- reported.
  4. History of unexplained fainting spells as self-reported.
  5. History of head injury resulting in more than a momentary loss of consciousness as self-reported.
  6. History of brain surgery as self-reported.
  7. Suffering from severe depression.
  8. Active malignancy.

For age-matched controls:

1. Recently started on antiepileptic drug therapy.
2. History of neurological disorders involving stroke, brain tumors, or epilepsy as self- reported.
3. History of unexplained fainting spells as self-reported.
4. History of head injury resulting in more than a momentary loss of consciousness as self-reported.
5. History of brain surgery as self-reported.
6. Suffering from severe depression.
7. Active malignancy.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 22-85 years who live locally and consent will be enrolled in two groups: an OUD cohort (DSM-5 opioid use disorder ≥6 months, positive urine toxicology, ongoing craving) and an age-matched non-OUD control group. All must reside in the study area with no relocation plans. Exclusion criteria (both cohorts) include recent antiepileptic initiation; history of stroke, brain tumor, epilepsy, unexplained syncope, significant head injury with loss of consciousness, or brain surgery; severe depression; active malignancy; and, for OUD subjects, recent ingestion of poppy seeds or Papaveris fructus products.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Electroencephalogram power in Delta through Gamma bands | 1 week
  High-density electroencephalogram power will be assessed during rest (eyes open, eyes closed) and activity

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical & Imaging Research Outcomes Lab, Chicago, Illinois, United States